CLINICAL TRIAL: NCT06580613
Title: Sustainable Hypertension Management in Primary Health Care in Sweden - Ett hållbart omhändertagande av Blodtryckspatienter i primärvården
Brief Title: Sustainable Hypertension Management in Primary Health Care in Sweden
Acronym: SHIP-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-03625-01
Record Dates: First submitted 2024-08-21; First posted 2024-08-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: Primary Health Care; Management
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): At the Control Primary Health Care Centers care continues as usual
  Interventions: Other: Control
- Intervention (Experimental): Hypertension management based on cardiovascular risk assessment. Low/medium risk: Digital contact with nurse, contact with GP only if needed High risk: Planned contacts with GP Group education on Hypertension for staff and participants
  Interventions: Other: New model of Hypertension Management

INTERVENTIONS:
Other: New model of Hypertension Management — Hypertension management based on cardiovascular risk assessment. For details see description of study arm intervention.
  Arms: Intervention
Other: Control — Hypertension Management as usual
  Arms: Control

SUMMARY:
New sustainable models of patient-focused and team-based care for patients with hypertension should be developed to achieve health improvements and cost-efficiency.

The aim of this project is to evaluate new ways of sustainable hypertension (HT) management in primary care, starting with a pilot study at 2 Primary Health Care Centres (PHCCs).

At intervention PHCCs cardiovascular risk is assessed with SCORE2 for all hypertension patients. The staff receives education on HT treatment and an easy-to-follow treatment protocol. Non-physicians lead patient education on HT in groups. Patients receive a home blood pressure (BP) monitor and communicate digitally with the assigned nurse on medication update, blood and urinary tests and follow up. The nurse consults with the physician if needed. Regular face to face visits with the physician are only scheduled for patients with high cardiovascular risk or end organ damage, otherwise for all patients if needed.

At the control PHCs hypertension care continues as usual. All participants will be asked to complete questionnaires after 6 and 24 months.

Outcomes are feasibility for the pilot study and the proportion of patients reaching BP target plus change in systolic BP, cardiovascular risk factors, patients´ and staff´s grade of satisfaction and knowledge, and health care costs for the main study, compared between intervention and control PHCCS. Results will help to establish sustainable models of treating HT patients in Primary Care.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients with hypertension

Exclusion Criteria:

* secondary hypertension according to the medical records at the Primary Health Care Center
* terminal illness
* pregnancy-induced hypertension
* cognitive impairment
* impaired vision (not able to read measurements for the home BP measurements or communicate via "1177 direct" digitally)
* psychotic disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure change | 6 months
  change in proportion of patients reaching blood pressure target of <140/90 mmHg
Blood pressure change | 24 months
  change in proportion of patients reaching blood pressure target of <140/90 mmHg

SECONDARY OUTCOMES:
Health economic evaluation | 24 months
  Estimation of the ICER values (cost per unit of effect). Calculation of QALY, based on EQ5D (questionnaires). Comparison of ICER per QALY with values from the National Board of Health and Welfare
Participants grade of satisfaction | 24 months
  Questionnaires. 7 point Likert Scale: Level of Satisfaction - 7 point
  1. - Completely dissatisfied
  2. - Mostly dissatisfied
  3. - Somewhat dissatisfied
  4. - neither satisfied or dissatisfied
  5. - Somewhat satisfied
  6. - Mostly satisfied
  7. - Completely satisfied
Staffs grade of satisfaction | 24 months
  Questionnaires. 7 point Likert Scale: Level of Satisfaction - 7 point
  1. - Completely dissatisfied
  2. - Mostly dissatisfied
  3. - Somewhat dissatisfied
  4. - neither satisfied or dissatisfied
  5. - Somewhat satisfied
  6. - Mostly satisfied
  7. - Completely satisfied
Blood glucose level and cholesterol | 24 months
  Change in mean blood glucose level (mmol/l), mean LDL-cholesterol (mmol/l), mean HDL-cholesterol (mmol/l)
Kidney function | 24 months
  Change in mean eGFR (ml/min/1,73 m2)
Kidney complications | 24 months
  Change in % of patients with microalbuminuria (U-albumin/kreatinin-kvot (mg/mmol) 3,0-30)
Smoking | 24 months
  Change in % of patients who smoke)

CONTACTS AND LOCATIONS:
Locations (1):
- Husensjö Primary Health Care Center, Helsingborg, Sweden

IPD SHARING:
Plan to Share IPD: No